CLINICAL TRIAL: NCT07110987
Title: A Prospective Open-label Randomized Controlled Trial , Evaluating the Efficacy of Ursodeoxycholic Acid (UDCA) as an Adjuvant to Phototherapy in Neonates With Indirect Hyperbilirubinemia
Brief Title: The Efficacy of Ursodeoxycholic Acid (UDCA) as Adjuvant Therapy to Phototherapy in the Management of Neonatal Indirect Hyperbilirubinemia
Acronym: UDCA-Neo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tishreen University Hospital (Other)
Responsible Party: Principal Investigator, Ashraf Maan Alshelly, MD, Pediatric Resident, Tishreen University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Alshelly-UDCA-2025
Record Dates: First submitted 2025-07-13; First posted 2025-08-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Hyperbilirubinemia, Neonatal Indirect
Keywords: Neonatal Jundice; Phototherapy; Ursodeoxycholic acid; UDCA; G6pd Deficiency; Rh incompatibilty; ABO incompatibility; Adjuvant therapy
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Glucosephosphate Dehydrogenase Deficiency | interventions — Phototherapy; Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - phototherapy only (Active Comparator): Infants who have indirect hyperbilirubinemia recieve continuous triple phototherapy only .
  Interventions: Procedure: Phototherapy
- Group B - phototherapy + UDCA (Experimental): Phototherapy + UDCA
  Interventions: Procedure: Phototherapy; Drug: ursodeoxycholic acid (UDCA)

INTERVENTIONS:
Procedure: Phototherapy — Triple continuous phototherapy per AAP Guudelines
  Other Names: Triple continuous phototherapy
Drug: ursodeoxycholic acid (UDCA) — 10mg/kg/day orally divided in two doses (URSORASHA) . Given with feeds untill the bilirubin level drop down to limits that don't need therapy due to AAP guidelines.
  Other Names: Ursodiol; UDCA
  Arms: Group B - phototherapy + UDCA

SUMMARY:
This is a prospective, open-label, randomized controlled trial conducted at Lattakia University Hospital (Tishreen University), aiming to evaluate the efficacy of Ursodeoxycholic Acid (UDCA) as an adjuvant to triple phototherapy in the management of indirect hyperbilirubinemia in neonates ≥34 weeks of gestation.

Eligible neonates will be randomly assigned to one of two groups:

Group A: continuous triple phototherapy only

Group B: UDCA (10 mg/kg/day in two oral doses) in addition to triple continuous phototherapy.

Stratified randomization will be applied according to etiology (hemolytic, non-hemolytic, G6PD deficiency). The primary outcome is the rate and time of decline in total and indirect serum bilirubin to below phototherapy thresholds, monitored every 12 hours until discharge.

This trial seeks to determine whether UDCA may reduce phototherapy duration or enhance bilirubin clearance in a safe and effective manner.

Although this is an open-label trial for care providers and participants , the statstican conducting data analysis will be blinded to group allocation to reduce assessment bias.

DETAILED DESCRIPTION:
This is a prospective, open-label, randomized controlled clinical trial designed to assess the efficacy of ursodeoxycholic acid (UDCA) as an adjuvant to continuous triple phototherapy in neonates with indirect hyperbilirubinemia.

The study includes neonates ≥34 weeks gestational age and appropriate for gestational age (AGA), who meet the American Academy of Pediatrics (AAP) criteria for starting phototherapy.

Participants will be randomized 1:1 into two parallel arms:

Group A (Control): Continuous triple phototherapy

Group B (Intervention): Continuous triple phototherapy + oral UDCA at a dose of 10 mg/kg/day divided into two doses, using locally available Ursorasha (Rasha Pharma, license #1991/1192).

Randomization will be performed using stratified block randomization, with three stratification layers to balance known confounding factors across groups:

1. Hemolytic jaundice (ABO or Rh incompatibility)
2. Non-hemolytic jaundice (physiological or breast milk)
3. G6PD deficiency

Total serum bilirubin (TSB) will be monitored every 12 hours and compared across groups. Primary outcome is the time needed for bilirubin to drop below phototherapy threshold, according to age-specific AAP phototherapy nomograms.

Additional secondary analyses will include the rate of bilirubin decline at 24 and 48 hours, need for rescue therapy, and subgroup analysis based on gestational age (late preterm vs term), and jaundice type.

Based on retrospective hospital data, the anticipated enrollment is 70 neonates. However, due to the lower prevalence of G6PD deficiency, this subgroup may not yield enough cases for statistically powered subgroup analysis. It will instead be analyzed descriptively or as exploratory.

The study includes clearly defined inclusion/exclusion criteria and a unified therapeutic protocol applied to all infants.

Inclusion criteria: Neonates ≥34 weeks GA, AGA, with indirect hyperbilirubinemia requiring phototherapy.

Exclusion criteria: Neonates <34 weeks, non-AGA, suspected/confirmed sepsis, TPN, liver disorders, or infants of diabetic mothers.

This protocol was initiated and registered within 21 days of enrolling the first patient. The study has received initial approval from the Department of Pediatrics at Lattakia University Hospital (formerly Tishreen University Hospital) under Committee Decision #70. Final administrative ethics approval from the university is in progress due to procedural delays in our country.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates with gestational age ≥ 34 weeks
2. Appropriate for Gestational Age (AGA) infants
3. Presence of indirect hyperbilirubinemia that meets the threshold for phototherapy.

Exclusion Criteria:

1. Gestational age < 34 weeks
2. Small or Large for Gestational Age
3. Direct (conjugated) hyperbilirubinemia > 20% of total bilirubin
4. Suspected or confirmed sepsis
5. Neonates of diabetic mothers
6. Presence of congenital or acquired liver disease
7. Receiving Total Parenteral Nutrition (TPN)

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of total serum bilirubin to below phototherapy threshold | Day 0 to Day 7
  Measurement of serum total bilirubin levels every 12 hours until they fall below the phototherapy threshold based on gestational age and postnatal age. Outcome is considered achieved once bilirubin levels drop below threshold and phototherapy can be discontinued .
Time to bilirubin reduction below treatment threshold | Day 0 to Day 7
  Time (in hours) from treatment initiation to TSB falling below phototherapy threshold in each group.
Mean reduction in total serum bilirubin at 12 hours | 12 hours of starting therapy
  To compare the average decrease in total serum bilirubin after 12 hours between the two groups.

SECONDARY OUTCOMES:
Comparison of Hospital stay between both groups | Day 0 to Day 7
  The total length of hospital stay (in days) will be compared between both groups (phototherapy alone and UDCA + phototherapy) to assess the impac5 of UDCA on hospital stay duration.
Comparison of bilirubin reduction between late preterm (34weeks-36weeks+6 days) and term infants (≥37 weeks) in each treatment group. | Up to 7 Days
  This outcome aims to evaluate whether the gestational maturity of neonates affects the response to the assigned treatment. The kinetics of bilirubin reduction (mg/dL over time) will be analyzed separately within the phototherapy-only group and the phototherapy + UDCA group, comparing late preterm and term neonates.
Comparison of bilirubin decline in each gestational age group (preterm vs preterm) and (term vs term) across jaundice types between treatment arms. | Day 0 to Day 7.
  This outcome investigates whether the effectiveness of UDCA as an adjuvant varies by both gestational age and jaundice type. Within each gestational age group (late preterm and term), the bilirubin decline trends in rate (mg/dl) will be compared between the treatment groups across each of the following etiologies:
  * Hemolytic jaundice
  * Non-hemolytic jaundice
  * G6PD-related jaundice
Need for retreatment | Day 0 to Day 10 , Up to 3 days after treatment discontinuation.
  percentage of infants who required re-initiation of phototherapy after initial discontinuation in each Arm .
Incidence of adverse effects in the UDCA group | Day 0 to Day 7
  Any reported side effects in neonates receiving UDCA
Time to bilirubin reduction below threshold between treatment groups within each gestational age category | Up to 7 Days
  Time from initiation of treatment to bilirubin falling below treatment threshold for:
  * Late preterm (34-36+6 weeks): Group A vs. Group B
  * Term (≥37 weeks): Group A vs. Group B
Time to bilirubin reduction between late preterm and term neonates within each treatment group | Up to 7 Days
  To assess whether gestational age affects time to bilirubin normalization within each group.
Time to bilirubin normalization in each gestational age group across jaundice types | Up to 7 Days.
  For each gestational age (late preterm, term), compare time to normalization among jaundice types (hemolytic, non-hemolytic, G6PD) between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan H Dayoub, Prof.Neonat, Study Director — Lattakia university hospital (Tishreen university Hospital ) , Lattakia university
Locations (1):
- Lattakia University Hospital, Latakia, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodrigues CM, Steer CJ. The therapeutic effects of ursodeoxycholic acid as an anti-apoptotic agent. Expert Opin Investig Drugs. 2001 Jul;10(7):1243-53. doi: 10.1517/13543784.10.7.1243. PMID 11772248
- [Result] 2. Wang H, et al. Effect of ursodeoxycholic acid on neonatal indirect hyperbilirubinemia: A meta-analysis. World J Pediatr. 2022;18(5):375-383. PMID: 35689782
- [Result] 3. Hassan NM, El Said NM. Role of ursodeoxycholic acid in treatment of neonatal indirect hyperbilirubinemia. Iraqi J Pediatr. 2015;32(1):42-47.
- [Result] Ughasoro MD, Adimorah GN, Chukwudi NK, Nnakenyi ID, Iloh KK, Udemba CE. Reductive effect of ursodeoxycholic acid on bilirubin levels in neonates on phototherapy. Clin Exp Gastroenterol. 2019 Jul 29;12:349-354. doi: 10.2147/CEG.S207523. eCollection 2019. PMID 31534356
- [Result] Rezaie M, Gholami R, Jafari M, Haghighinejad H. Evaluating the effect of ursodeoxycholic acid on total bilirubin of neonates with glucose-6-phosphate dehydrogenase deficiency complicated by indirect hyperbilirubinaemia. J Paediatr Child Health. 2021 Aug;57(8):1175-1181. doi: 10.1111/jpc.15411. Epub 2021 Mar 8. PMID 33682983
- See also: PubMed - Meta-analysis on UDCA in neonates — https://pubmed.ncbi.nlm.nih.gov/35689782/